CLINICAL TRIAL: NCT00639158
Title: A Multicenter, Randomized, Double-Blind, Prospective Study Comparing the Safety and Efficacy of ABT-335 in Combination With Atorvastatin and Ezetimibe to Atorvastatin in Combination With Ezetimibe in Subjects With Combined (Atherogenic) Dyslipidemia
Brief Title: Safety and Efficacy Study Comparing ABT-335 Coadministered With Atorvastatin and Ezetimibe to Atorvastatin Coadministered With Ezetimibe in Subjects With Multiple Abnormal Lipid (Fat) Levels in the Blood
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Maureen Kelly, MD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-275
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Results first posted 2009-11-05 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2011-06

CONDITIONS: Dyslipidemias; Coronary Heart Disease; Combined (Atherogenic) Dyslipidemia; Mixed Dyslipidemia
MeSH Terms: conditions — Dyslipidemias; Coronary Disease | interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; Fenofibrate; fenofibric acid; Atorvastatin; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABT-335 + atorvastatin + ezetimibe (Active Comparator)
  Interventions: Drug: ABT-335; Drug: atorvastatin; Drug: ezetimibe
- Placebo + atorvastatin + ezetimibe (Placebo Comparator)
  Interventions: Drug: placebo; Drug: atorvastatin; Drug: ezetimibe

INTERVENTIONS:
Drug: ABT-335 — 135 mg capsule, daily, 12 weeks
  Other Names: TriLipix; Fenofibric acid; Choline Fenofibrate
  Arms: ABT-335 + atorvastatin + ezetimibe
Drug: placebo — placebo capsule, daily, 12 weeks
  Arms: Placebo + atorvastatin + ezetimibe
Drug: atorvastatin — 40 mg, tablet, daily, 12 weeks
  Other Names: Lipitor
Drug: ezetimibe — 10 mg capsule, daily, 12 weeks
  Other Names: Ezetrol; Zetia; Ezemibe

SUMMARY:
The primary purpose of this study is to compare the safety and efficacy of ABT-335 (investigational drug) coadministered with atorvastatin and ezetimibe to atorvastatin coadministered with ezetimibe in subjects with abnormal lipid (fat) levels in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mixed dyslipidemia (trigylcerides, > or = to 150 mg/dL to < 400 mg/dL; HDL-C < 40 mg/dL for males, < 50 mg/dL for females; LDL-C, > or = to 130 mg/dL).
* Subjects must agree to use adequate birth control methods and to adhere to the American Heart Association (AHA) Diet.

Exclusion Criteria:

* Subjects with unstable or uncontrolled medical conditions considered inappropriate in a clinical trial.
* Subjects with an unstable dose of medications or receiving Coumadin, oral, intravenous or intramuscular cyclosporine, statins, or certain other medications.
* Women who are pregnant or plan on becoming pregnant, or women who are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (110):
- United States (110):
  - Birmingham, Alabama
  - Columbiana, Alabama
  - Hueytown, Alabama
  - Ozark, Alabama
  - Tuscaloosa, Alabama
  - Sierra Vista, Arizona
  - Hot Springs, Arkansas
  - Carmichael, California
  - Concord, California
  - Long Beach, California
  - Los Angeles, California
  - Norwalk, California
  - Roseville, California
  - Sacramento, California
  - Santa Ana, California
  - Tustin, California
  - West Hills, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Clearwater, Florida
  - Delray Beach, Florida
  - Fort Myers, Florida
  - Holly Hill, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Longwood, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - New Smyrna Beach, Florida
  - Ocala, Florida
  - Ormond Beach, Florida
  - Pembroke Pines, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Roswell, Georgia
  - Suwanee, Georgia
  - Woodstock, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Peoria, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Arkansas City, Kansas
  - Overland Park, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Mount Sterling, Kentucky
  - Slidell, Louisiana
  - Baltimore, Maryland
  - Oxon Hill, Maryland
  - Brockton, Massachusetts
  - Edina, Minnesota
  - Olive Branch, Mississippi
  - City of Saint Peters, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Elizabeth, New Jersey
  - Hillsborough, New Jersey
  - Trenton, New Jersey
  - Johnson City, New York
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Morehead City, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Mason, Ohio
  - Mogadore, Ohio
  - Warren, Ohio
  - Tulsa, Oklahoma
  - Hillsboro, Oregon
  - Duncansville, Pennsylvania
  - Harleysville, Pennsylvania
  - Jersey Shore, Pennsylvania
  - Lansdale, Pennsylvania
  - Melrose Park, Pennsylvania
  - Newtown, Pennsylvania
  - Perkasie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Tipton, Pennsylvania
  - Warminster, Pennsylvania
  - Cumberland, Rhode Island
  - Anderson, South Carolina
  - Greenville, South Carolina
  - Greer, South Carolina
  - Simpsonville, South Carolina
  - Summerville, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Roanoke, Virginia
  - Virginia Beach, Virginia
  - Spokane, Washington
  - Madison, Wisconsin

REFERENCES:
- [Derived] Jones PH, Goldberg AC, Knapp HR, Kelly MT, Setze CM, Stolzenbach JC, Sleep DJ. Efficacy and safety of fenofibric acid in combination with atorvastatin and ezetimibe in patients with mixed dyslipidemia. Am Heart J. 2010 Oct;160(4):759-66. doi: 10.1016/j.ahj.2010.06.045. PMID 20934572

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject was randomized to the atorvastatin and ezetimibe treatment group and never received study drug.
Period: Overall Study
Arm/Group | ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe | Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe
Started | 272 (All randomized subjects were treated.) | 270 (1 subject was randomized but not treated because of an abnormal ECG that precluded treatment.)
Completed | 246 (26 subjects prematurely discontinued treatment.) | 240 (30 subjects prematurely discontinued treatment)
Not Completed | 26 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe | Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe | Total
Number analyzed (Participants) | 272 | 270 | 542
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 227 | 206 | 433
  >=65 years | 45 | 64 | 109
Age Continuous [Mean (Standard Deviation); unit: years] | 54.4 (11.23) | 56.4 (10.67) | 55.4 (10.99)
Age Continuous [Mean (Standard Deviation); unit: participants]
  United States | 54.4 (11.23) | 56.4 (10.67) | 55.4 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 155 | 298
  Male | 129 | 115 | 244

OUTCOME MEASURES:

1. Primary Outcome: Median Percent Change in Triglycerides From Baseline to Final Visit
Description: [(Week 12 triglycerides minus baseline triglycerides)/baseline triglycerides] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline triglyceride value and at least 1 postbaseline triglyceride value, last observation carried forward.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe | Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe
Number analyzed (Participants) | 262 | 262
Percent change | -57.3 (22.32) [-67.1 to -46.3] | -39.7 (29.44) [-52.5 to -20.9]
Statistical Analysis 1: Comparison: ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe vs Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe; A sample size of 212 per arm provided 90% power and > 99% power with a 2-sided alpha = 0.05 level to detect differences between treatment arms of 6% and 17% in the percent change in HDL-C and TG, respectively, assuming an SD of 19% and 30%, respectively. This sample size provided an overall power of approximately 90% for the 2 primary comparisons. If a loss to follow-up rate of 8% was assumed, the sample size needed to be increased to 230 per arm to maintain the above power; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — The treatment group comparisons for both primary efficacy variables must have demonstrated superiority of ABT-335 + atorvastatin + ezetimibe to declare this arm successful. Thus, no adjustments were made for multiple comparisons

2. Secondary Outcome: Mean Percent Change in Apolipoprotein AI (apoAI) From Baseline to Final Visit
Description: [(Week 12 apoAI minus baseline apoAI)/baseline apoAI] x 100
Time Frame: Baseline to 12 weeks (Final Visit)
Population: All randomized subjects with a baseline apoAI value and at least 1 postbaseline apoAI value, last observation carried forward.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe | Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe
Number analyzed (Participants) | 248 | 239
Percent change | 1.8 (0.74) | -1.3 (0.76)
Statistical Analysis 1: Comparison: ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe vs Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe; Secondary endpoints were tested in fixed sequence. If superiority of ABT-335 + atorvastatin + ezetimibe treatment was demonstrated for primary endpoints, secondary endpoints were tested in ranked order of apoA1, VLDL-C, apoC3, non-HDL-C, apoB, and hsCRP at alpha = 0.05 level until 1 secondary endpoint failed to reach statistical significance; Test type: Superiority or Other; p = 0.004, ANCOVA; Corresponding baseline lipid value as the covariate and with effect for treatment group

3. Primary Outcome: Mean Percent Change in High-Density Lipoprotein Cholesterol (HDL-C) From Baseline to Final Visit
Description: [(Week 12 HDL-C minus baseline HDL-C)/baseline HDL-C] x 100
Time Frame: Baseline to 12 weeks (Final Visit)
Population: All randomized subjects with a baseline high density lipoprotein cholesterol (HDL-C) value and at least 1 postbaseline HDL-C value, last observation carried forward.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe | Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe
Number analyzed (Participants) | 262 | 262
Percent change | 13.0 (0.95) | 4.2 (0.95)
Statistical Analysis 1: Comparison: ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe vs Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Corresponding baseline lipid value as the covariate and with effect for treatment group

4. Secondary Outcome: Mean Percent Change in Very Low-Density Lipoprotein Cholesterol (VLDL-C) From Baseline to Final Visit
Description: [(Week 12 VLDL-C minus baseline VLDL-C)/baseline VLDL-C] x 100
Time Frame: Baseline to 12 weeks (final visit)
Population: All randomized subjects with a baseline VLDL-C value and at least 1 postbaseline VLDL-C value, last observation carried forward.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe | Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe
Number analyzed (Participants) | 261 | 262
Percent change | -57.8 (1.87) | -41.1 (1.87)
Statistical Analysis 1: Comparison: ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe vs Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Corresponding baseline lipid value as the covariate and with effect for treatment group

5. Secondary Outcome: Mean Percent Change in Apolipoprotein CIII (apoCIII) From Baseline to Final Visit
Description: [(Week 12 apoCIII minus baseline apoCIII)/baseline apoCIII] x 100
Time Frame: Baseline to 12 weeks (Final Visit)
Population: All randomized subjects with a baseline apoCIII value and at least 1 postbaseline apoCIII value, last observation carried forward.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe | Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe
Number analyzed (Participants) | 249 | 242
Percent change | -42.5 (1.22) | -25.3 (1.23)
Statistical Analysis 1: Comparison: ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe vs Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Corresponding lipid value as the covariate and with effect for treatment group

6. Secondary Outcome: Mean Percent Change in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) From Baseline to Final Visit
Description: [(Week 12 non-HDL-C minus baseline non-HDL-C)/baseline non-HDL-C] x 100
Time Frame: Baseline to 12 weeks (Final Visit)
Population: All randomized subjects with a baseline non-HDL-C value and at least 1 postbaseline non-HDL-C value, last observation carried forward.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe | Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe
Number analyzed (Participants) | 262 | 262
Percent change | -55.6 (0.94) | -51.0 (0.94)
Statistical Analysis 1: Comparison: ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe vs Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Corresponding baseline lipid value as the covariate and with effect for treatment group

7. Secondary Outcome: Mean Percent Change in Apolipoprotein B (apoB) From Baseline to Final Visit
Description: [(Week 12 apoB minus baseline apoB)/baseline apoB] x 100
Time Frame: Baseline to 12 weeks (Final Visit)
Population: All randomized subjects with a baseline apoB value and at least 1 postbaseline apoB value, last observation carried forward.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe | Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe
Number analyzed (Participants) | 248 | 239
Percent change | -49.1 (0.91) | -44.7 (0.93)
Statistical Analysis 1: Comparison: ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe vs Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Corresponding baseline lipid value as the covariate and with effect for treatment group

8. Secondary Outcome: Median Percent Change in High-Sensitivity C-Reactive Protein (hsCRP) From Baseline to Final Visit
Description: [(Week 12 hsCRP minus baseline hsCRP)/baseline hSCRP] x 100
Time Frame: Baseline to 12 weeks (Final Visit)
Population: All randomized subjects with a baseline hsCRP value and at least 1 postbaseline hsCRP value, last observation carried forward.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe | Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe
Number analyzed (Participants) | 261 | 262
Percent change | -52.1 (102.82) [-67.4 to -25.4] | -40.3 (516.56) [-60.6 to -13.4]
Statistical Analysis 1: Comparison: ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe vs Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Rank-sum test

ADVERSE EVENTS:
Arm/Group | ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe | Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe
Serious Adverse Events (participants affected / at risk) | 3/272 | 5/270
Other Adverse Events (participants affected / at risk) | 41/272 | 51/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe (N=272) | Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe (N=270)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Esophageal Pain (Gastrointestinal disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Wound Infection Staphylococcal (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-335 + 40 mg Atorvastatin + 10 mg Ezetimibe (N=272) | Placebo + 40 mg Atorvastatin + 10 mg Ezetimibe (N=270)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 10
Diarrhea (Gastrointestinal disorders) | 9 | 6
Fatigue (General disorders) | 6 | 10
Headache (Nervous system disorders) | 6 | 9
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 10 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 10
Nausea (Gastrointestinal disorders) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not to publish or present the results before the publication of the multi-center investigator paper, but in no event shall be so restricted after the expiration of twelve (12) months from completion of the studies at all sites. Any presentation or publication to be submitted to Sponsor (in Draft of the same) for Sponsor review and comment.